CLINICAL TRIAL: NCT04587648
Title: Cardiac Amyloidosis in Heart Failure Patients With Preserved Ejection Fraction
Brief Title: Cardiac Amyloidosis in HFpEF
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Jin-Shan branch (Unknown); National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 201906065RINA
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Amyloidosis Cardiac
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Sodium; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NA, observational study — NA, observational study

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) accounts for half of heart failure cases with heterogenous cause and variable presentations. The diagnosis of HFpEF required clinical signs and symptoms of HF, normal left ventricular ejection fraction (LVEF) and evidence of diastolic dysfunction. No treatment has been shown in recent major clinical trials having benefits in these patients. One major reason of the poor response to medical treatment is the heterogeneity of HFpEF, which contains many different underline causes. To identify the underlying causes of HFpEF may improve the diagnosis and treatment in these patients.

Age-related amyloid deposition has first been reported in 1876 and the following autopsy studies showed the prevalence of senile cardiac amyloid is up to 25%. Recently, it has been recognized that the deposits in senile cardiac amyloid are derived from wild-type transthyretin (TTR). Transthyretin amyloidosis cardiac amyloidosis (ATTR CA) is caused by myocardial deposition of misfolded transthyretin protein. There are 2 types of ATTR classified by genetic mutation including wild-type ATTR (ATTRwt) and familial cardiac amyloid caused by TTR mutation (ATTRm).

Multimodality techniques have been developed to assist in the diagnosis of the diagnosis of TTR. Among them, 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD) scintigraphy is a non-invasive test and it can diagnose TTR from other cause diverse form of cardiac amyloidosis and cardiomyopathy. In the study of Gonzalez-Lopez et al, in 120 HFpEF patients, 16 (13.3%) had positive 99mTc-DPD scan. Four patients with positive 99mTc-DPD scan received endomyocardial biopsy and confirmed cardiac amyloid deposition.

ATTRwt could be an important cause of HFpEF and it was often under diagnosed. A recent study in Spain reported that 13% of patents over age of 60 years with HFpEF and left ventricular wall thickness of 12mm or more had ATTRwt. However, the prevalence of ATTRwt among patients with HFpEF is not well-established in Taiwan and Asia. The aim of this study is to determine the prevalence, clinical characteristics, risk factors and outcomes of ATTRwt related HFpEF patients in Taiwan.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a heterogeneous clinical situation with multiple underlying causes. The diagnosis of HFpEF is challenging which requires clinical signs/symptoms of HF, a normal or mildly impaired systolic function measured by left ventricular ejection fraction (LVEF), and evidence of diastolic dysfunction. There are no significant improvements in treatment of HFpEF in recent years and the results in the major clinical trials for HFpEF were disappointed. One major reason is the heterogeneity of HFpEF, which contains several diseases under the same entity.

Small deposits of amyloid are found in the elder hearts in up to 25% of the autopsies. These deposits are mainly composed by wild-type transthyretin (TTR). Transthyretin amyloidosis cardiac amyloidosis (ATTR CA) is caused by myocardial deposition of misfolded transthyretin protein. It is classified into 2 groups by the genetics of Transthyretin amyloidosis (ATTR): wild-type (ATTRwt) or hereditary (hATTR or ATTRm). ATTR CA, irrespective of genotype, is an unrecognized mechanism underlying HFpEF. It was reported wild-type TTR might be an underdiagnosed cause of HFpEF. However, the prevalence of wild-type ATTR among patients with HFpEF is not well-established in Taiwan and Asia.

One of the most convenient method to detect and diagnosis cardiac amyloidosis is 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD) scintigraphy6. In the study of Gonzalez-Lopez et al, in 120 HFpEF patients, 16 (13.3%) had positive 99mTc-DPD scan6. Four patients with positive 99mTc-DPD scan received endomyocardial biopsy and confirmed cardiac amyloid deposition6. In addition, technetium-99m TC pyrophosphate (PYP) scintigraphy is also very useful in diagnosis of cardiac amyloidosis.

The propose of this study is to determine the prevalence of ATTRwt among elderly HFpEF patients in Taiwan. In this study, the investigators will recruit a cohort of HFpEF patients in Taiwan to define the number of patients who have cardiac amyloidosis by utilizing highly sensitive heart imaging and blood tests. The investigators will also explore differences in different risk factors as they relate to heart failure disease progression in cardiac amyloidosis. According our previous studies, the average age of HFpEF in Taiwan is 65 y/o. In this study, the investigators set age limitation as 60 y/o. However, because 5% ATTRwt were < 60 y/o9, therefore, the investigators also recruit patients >50y/o with risk factors of ATTRwt.

Hypothesis HFpEF is a heterogeneous clinical situation with multiple underlying causes. ATTRwt is an underdiagnosed cause of HFpEF but the prevalence is unknown in Taiwan. ATTRwt can be diagnosed non-invasively by 99mTc-PYP scintigraphy7. The investigators aimed to investigate the prevalence and clinical characteristics of ATTRwt among patients with HFpEF.

Primary Objective(s) / Endpoint(s) Percentage of participants with ATTRwt among patients with HFpEF in Taiwan

Secondary Objective(s) / Endpoint(s) To investigate the clinical and echocardiographic characters in ATTRwt patients and compare with HFpEF patients without ATTRwt

Trial Population Eligible HFpEF patients with a LVEF of ≧50%, New York Heart Association (NYHA) class I-IV symptoms: Both in-patients or patients in clinics could be enrolled. These patients could be newly diagnosed or has been diagnosed. Study subjects will be pre-stratified according to left ventricular posterior wall thickness (LVPW) ≥12mm or less; number of subjects with LVPW ≥12mm should account for more than 50% of total subjects recruited in the final analysis.

Sample Size and Sample Size Justification The study will prospectively evaluate the prevalence of ATTRwt among patients with HFpEF. Assume the expected 10% prevalence of ATTRwt in patients with HFpEF, the target recruitment of 260 HFpEF patients would yield 25 ATTRwt positive result, which would provide the prevalence estimate with associated 90% confidence interval at the range of +- 3%. The estimated enrolled time is 18 months.

Key Inclusion Criteria

1. Patient is ≥ 60 years old or 50 y/o with carpal tunnel syndrome or spinal stenosis
2. Patient has been diagnosed as HFpEF in their medical history or newly diagnosed as HFpEF. They have HF symptoms with NYHA Classification of I-IV when diagnosis. The criteria of HFpEF is according to our previous studies10.
3. More than 50% of them have LVPW ≥12mm (when diagnosis).
4. Written informed consent could be obtained

Key Exclusion Criteria

1. Patients unwilling to join this projects
2. Patients with unstable coronary artery disease, plan to receive coronary intervention within months.
3. Patients has previous history of heart failure reduced ejection (HFrEF) with a LVEF <40%.

Method

1. Patients recruitment and study protocol The enrolled and exclusion criteria were mentioned above. The investigators will enroll 260 HFpEF patients (> 50% with LVPW thickness >12mm). After receiving informed consent, patients will receive NTproBNP, ECG, and echocardiography. Then the investigators will arrange 99mTc-PYP scan to detect the presence of amyloidosis. If patients have these data (ECG, NTproBNP, echocardiogram, 99mTc PYP) within 6 months, the investigators will record and use this data and do not perform again. In patients with positive 99mTc-PYP scan, the investigators will detect urinary monoclonal light chain and serum monoclonal light chain. In addition, the investigators will arrange TTR genetic testing.
2. Data Collection Delegated physicians or study personnel blinded to scintigraphy results will review the medical records of all patients. Demographic and clinical data will be collected during outpatient clinic visit.
3. Scintigraphy Protocol Planar and single-photon positive emission computed tomography (SPECT) imaging with 99mTc-PYP was performed with a dual head Philips Precedence SPECT/CT camera (Philips Healthcare, Guildford, United Kingdom). Patients received 20 to 25 mCi of 99mTc-PYP intravenously and images were obtained at 2 hours over 8 minutes duration.
4. Genotype Testing The TTR mutation was confirmed by sequencing of the TTR gene following National Taiwan University Hospital established protocols. All 4 exons and their flanking intron regions of the human TTR gene were amplified by polymerase chain reaction (PCR). The amplicons were purified by the Gel/PCR DNA Fragments Extraction Kit (Geneaid, Taipei, Taiwan). Sequencing was performed at the corresponding exons by using the ABI3730 automatic DNA sequencer (Applied Biosystems, Foster City, CA).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 60 years old or 50 y/o with carpal tunnel syndrome or spinal stenosis
* Patient has been diagnosed as HFpEF in their medical history or newly diagnosed as HFpEF. They have HF symptoms with NYHA Classification of I-IV when diagnosis. The criteria of HFpEF is according to our previous studies.
* More than 50% of them have LVPW ≥12mm (when diagnosis).
* Written informed consent could be obtained.

Exclusion Criteria:

* Patients unwilling to join this projects.
* Patients with unstable coronary artery disease, plan to receive coronary intervention within months.
* Patients has previous history of HFrEF with a LVEF <40%.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible HFpEF patients with a LVEF ≥50%, NYHA class I-IV symptoms: Both in-patients or patients in clinics could be enrolled. These patients could be newly diagnosed or has been diagnosed. Study subjects will be pre-stratified according to left ventricular posterior wall thickness (LVPW) ≥12mm or less; number of subjects with LVPW ≥12mm should account for more than 50% of total subjects recruited in the final analysis.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ATTRwt among patients with HFpEF in Taiwan | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided